CLINICAL TRIAL: NCT06201624
Title: Oral Isotretinoin in The Treatment of Melasma A Randomized Controlled Clinical Trial
Brief Title: Oral Isotretinoin in Melasma a Randomized Controlled Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hagar Nofal, Lecturer of Dermatology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZU-IRB#10462/26-2-2023
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Isotretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isotretinoin (Experimental): patients will receive oral isotretinoin (1 mg/kg/day) for 3 months
  Interventions: Drug: Isotretinoin
- Kligman Formula arm (Active Comparator): patients will receive topical triple combination formula at night everyday over the affected areas for 3 months
  Interventions: Drug: Triple combination formula

INTERVENTIONS:
Drug: Isotretinoin — Patients will receive 1mg/kg/day for 3 months
  Arms: Isotretinoin
Drug: Triple combination formula — Patients are instructed to apply the triple combination formula at night daily for 3 months
  Other Names: modified Kligman formula
  Arms: Kligman Formula arm

SUMMARY:
Melasma is a common refractory acquired hyperpigmentation of the skin having a serious impact on patients' quality of life. Melasma is challenging to treat. Treatment is often a multimodality approach. Due to the attached psychological and social stress, it is important to counsel patients with melasma adequately about the chronicity of the disease, the importance of photoprotection, and the role of hormones in disease persistence before embarking on therapeutic correction. So in this study, we are exploring the efficacy of oral isotretinoin for treating melasma.

DETAILED DESCRIPTION:
Melasma has a significant impact on the quality of life and self-esteem of those affected. Darker skin photo types e.g. Egyptians have excess potential to develop melasma.

Melasma is a chronic and challenging condition to manage. Previous treatment modalities have been unsatisfactory.

Oral isotretinoin is a potential treatment modality for melasma that has not been investigated yet.

In this study we aim to evaluate the efficacy and the tolerability of oral isotretinoin in the treatment of melasma and to compare its efficacy and tolerability with the current gold standard "topical triple combination formula"

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years
2. Patients complaining of melasma.
3. Patients with all types of melasma (epidermal, dermal and mixed)
4. Sexually active women who is willing to follow at least 2 types of contraceptive methods during study period
5. Patients with skin type I-V

Exclusion Criteria:

1. Pregnant or nursing women.
2. Women on any concurrent therapy for melasma.
3. Patients that are using any therapy for melasma for the last 45 days.
4. Patient with abnormal liver function test or lipid profile.
5. Patients with allergy or hypersensitivity to the assigned drugs.
6. Women not willing to follow contraceptive methods at time of study.
7. Patients on facial treatments or photosensitizing drugs within previous 6 months.
8. Patients with back or joint pain.
9. Patients with pre-existing or dormant dermatologic disease on the face that could interfere with the outcome of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | three months
  Treatment efficacy will be assessed by the change in disease severity measured in mMASI at the end of the treatment period, and the difference in the global appearance of melasma through standardized photographs using Global Aesthetic Improvement Scale (GAIS) using a five-point ordinal scale (1 = exceptionally improved appearance, 2 = very improved appearance, 3 = improved appearance, 4 = unaltered appearance, 5 = worsened appearance). The duration taken till complete clearance will be assessed as well.
Time to complete clearance | 12 weeks
  The duration taken till complete clearance will be assessed as well.

SECONDARY OUTCOMES:
Quality of life index | 12 weeks
  The change in patients' quality of life using the difference between results of "Melasma Quality of Life Index" at baseline and end of treatment.
Treatment tolerability | 12 weeks
  Treatment tolerability will be assessed in terms of the side effects reported by the investigator or the patients in follow-up visits including but not limited to; facial erythema, scaling, a burning sensation, and cheilitis. Patients' compliance assessed by the percentage of patients withdraw from each arm of the study and the number of days per week the patients' take/apply their medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology department, Zagazig University Hospitals, Faculty of Medicine, Zagazig University, Zagazig, Select Region, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and a copy of the master sheet for data collection, the statistical analysis plan will be shared and the results will be published in a respective journal
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Artzi O, Horovitz T, Bar-Ilan E, Shehadeh W, Koren A, Zusmanovitch L, Mehrabi JN, Salameh F, Isman Nelkenbaum G, Zur E, Sprecher E, Mashiah J. The pathogenesis of melasma and implications for treatment. J Cosmet Dermatol. 2021 Nov;20(11):3432-3445. doi: 10.1111/jocd.14382. Epub 2021 Aug 19. PMID 34411403
- [Background] Garner ML, McShane DB, Burkhart CN, Morrell DS. Isotretinoin and vitiligo: can chronic cheilitis cause koebnerization? Pediatr Dermatol. 2015 May-Jun;32(3):e108-9. doi: 10.1111/pde.12538. Epub 2015 Mar 17. PMID 25781892
- [Background] Muthu SK, Narang T, Saikia UN, Kanwar AJ, Parsad D, Dogra S. Low-dose oral isotretinoin therapy in lichen planus pigmentosus: an open-label non-randomized prospective pilot study. Int J Dermatol. 2016 Sep;55(9):1048-54. doi: 10.1111/ijd.13293. Epub 2016 Apr 7. PMID 27062273